CLINICAL TRIAL: NCT04322942
Title: Comparison of the Diagnostic Accuracy of Monocyte Distribution Width and Procalcitonin on Sepsis in the Emergency Department
Brief Title: Sepsis Prediction by Monocyte Distribution Width and Procalcitonin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XPRPG3J0051
Record Dates: First submitted 2020-03-22; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Sepsis; Diagnoses Disease
Keywords: sepsis; procalcitonin; MDW
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (4):
- Non-infection
  Interventions: Diagnostic Test: Monocyte Distribution Width
- Infection without sepsis
  Interventions: Diagnostic Test: Monocyte Distribution Width
- Sepsis-2
  Interventions: Diagnostic Test: Monocyte Distribution Width
- Sepsis-3
  Interventions: Diagnostic Test: Monocyte Distribution Width

INTERVENTIONS:
Diagnostic Test: Monocyte Distribution Width — Monocyte Distribution Width as part of the CBC result.

SUMMARY:
The mortality rate of sepsis remains as high as 30 to 40%. Early diagnosis and treatment of patients with sepsis reduce mortality significantly. The most commonly used biomarkers in clinical practice are C-reactive protein (CRP) and procalcitonin (PCT). In terms of exploring new diagnostic tools of sepsis, monocyte distribution width (MDW) was first reported in 2017. It was reported as part of the white blood cell (WBC) differential count. MDW greater than 20 and abnormal WBC count together were reported to provide a satisfactory accuracy. The area under curve (AUC) in predicting sepsis-2 is 0.852. It was proposed as a novel diagnostic tool of sepsis in the emergency setting. Nonetheless, the performance of MDW compared with the conventional biomarkers remained unknown. The aim of this study was to compare the diagnostic accuracy of MDW and PCT on sepsis in the emergency department.

ELIGIBILITY:
Subject Inclusion Criteria

* Adult ≥20 years) subjects presenting to the ED with the chief complaints of fever, altered consciousness, hypotension, and dyspnea. CBC with differential testing performed, at presentation as part of their standard medical care.
* Subjects who have signed Informed Consent.

Subject Exclusion Criteria

* Previously enrolled in this study (i.e. subjects may not be enrolled more than once in this study)
* Subjects discharged from the ED <72 hours
* Pregnant women
* Subjects not able to understand or sign Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on a target of 75% sensitivity and lower limit of 65%, a minimum of 63 (will target 100) septic patients would be required. Higher numbers may be enrolled in the study to ensure adequate representation of sepsis cases. Given the estimated prevalence of the disease in the emergency department population (5-10%%), the number of non-septic patients is predicted to be significantly higher than septic. Based on the estimated prevalence of subjects who present and have blood draw, a minimum of 100 non-septic cases will be collected.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of predicting sepsis and sepsis-3 patients | within 2 hours after patient arrived ED.
  MDW, PCT, and other laboratory tests were all obtained at the same time with 2 hours after the patient was admitted to the emergency department (ED). Sensitivity and specificity of different cutoff value were calculated. Best cutoff value will be decided by the perfomance.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-huang Li, MD, Principal Investigator — Chang Gung Memorial Hospital, Linkou Medical Center
Locations (1):
- Chang Gung Memorial Hospital, Linkou Medical Center, Taoyuan District, 新北市, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li CH, Seak CJ, Chaou CH, Su TH, Gao SY, Chien CY, Ng CJ. Comparison of the diagnostic accuracy of monocyte distribution width and procalcitonin in sepsis cases in the emergency department: a prospective cohort study. BMC Infect Dis. 2022 Jan 4;22(1):26. doi: 10.1186/s12879-021-06999-4. PMID 34983430